CLINICAL TRIAL: NCT00691093
Title: Observational Study In Patients With Overactive Bladder (OAB) Treated With Toviaz® After Failure Of Previous Antimuscarinic Therapy Due To Ineffectivity Or Intolerance.
Brief Title: Study In Patients With Overactive Bladder Treated With Toviaz® After Failure Of Previous Therapy
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0221059
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Overactive Bladder; Urinary Incontinence
Keywords: observational
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — fesoterodine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fesoterodine
  Interventions: Drug: fesoterodine

INTERVENTIONS:
Drug: fesoterodine — 4 mg per 24 hours, possibility to increase to 8 mg depending on efficacy chronic treatment
  Other Names: TOVIAZ

SUMMARY:
This is a observational study in patients treated with fesoterodine (Toviaz), who have failed on previous treatment for overactive bladder. It will collect epidemiological data and investigate the efficacy and tolerability of fesoterodine.

DETAILED DESCRIPTION:
patients older than 18 years with overactive bladder after failure of previous antimuscarinic therapy (due to lack of efficacy or intolerance)

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with OAB after failure of previous antimuscarinic therapy - due to lack of efficacy: persistence of storage symptoms.
* Required symptoms: micturition frequency 8 and more / 24 hours and urgency episodes ≥2 per day subjectively perceived as bothersome
* Due to intolerance: persistent and/or unacceptable adverse events

Exclusion Criteria:

* Hypersensitivity to the active substance or to peanut or soya or any of the excipients.
* History of acute urinary retention (requiring catheterisation)
* Gastric retention
* Uncontrolled narrow angle glaucoma
* Myasthenia gravis
* Severe hepatic impairment (Child Pugh C)
* Concomitant use of potent CYP3A4 inhibitors in subjects with moderate to severe hepatic or renal impairment
* Severe ulcerative colitis
* Toxic megacolon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients older than 18 years with overactive bladder after failure of previous antimuscarinic therapy (due to lack of efficacy or intolerance)
Sampling Method: Non-Probability Sample
Enrollment: 823 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- Slovakia (54):
  - Pfizer Investigational Site, ?a?a
  - Pfizer Investigational Site, Aa
  - Pfizer Investigational Site, Adca
  - Pfizer Investigational Site, B.Bystrica
  - Pfizer Investigational Site, Banská Bystrica
  - Pfizer Investigational Site, Bardejov
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Dolný Kubín
  - Pfizer Investigational Site, Dunajská Streda
  - Pfizer Investigational Site, Hlohovec
  - Pfizer Investigational Site, Humenné
  - Pfizer Investigational Site, Ilina
  - Pfizer Investigational Site, Koice-aca
  - Pfizer Investigational Site, Koice
  - Pfizer Investigational Site, Komárno
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Kraovsky Chlmec
  - Pfizer Investigational Site, Liptovský Hrádok
  - Pfizer Investigational Site, Liptovský Mikuláš
  - Pfizer Investigational Site, Luenec
  - Pfizer Investigational Site, Malacky
  - Pfizer Investigational Site, Martin
  - Pfizer Investigational Site, Michalovce
  - Pfizer Investigational Site, Myjava
  - Pfizer Investigational Site, Námestovo
  - Pfizer Investigational Site, Nitra
  - Pfizer Investigational Site, Nové Zámky
  - Pfizer Investigational Site, Piešťany
  - Pfizer Investigational Site, Poprad
  - Pfizer Investigational Site, Povaska Bystrica
  - Pfizer Investigational Site, Považská Bystrica
  - Pfizer Investigational Site, Preov
  - Pfizer Investigational Site, Prievidza
  - Pfizer Investigational Site, Púchov
  - Pfizer Investigational Site, Revúca
  - Pfizer Investigational Site, Rimavská Sobota
  - Pfizer Investigational Site, Ruomberok
  - Pfizer Investigational Site, Ružomberok
  - Pfizer Investigational Site, Senica
  - Pfizer Investigational Site, Skalica
  - Pfizer Investigational Site, Sobrance
  - Pfizer Investigational Site, SpisskaNova Ves
  - Pfizer Investigational Site, Stropkov
  - Pfizer Investigational Site, Svidník
  - Pfizer Investigational Site, Topoany
  - Pfizer Investigational Site, Trebišov
  - Pfizer Investigational Site, Trenčín
  - Pfizer Investigational Site, Trenin
  - Pfizer Investigational Site, Trnava
  - Pfizer Investigational Site, Turianske Teplice
  - Pfizer Investigational Site, Urany
  - Pfizer Investigational Site, Vranov n/Topou
  - Pfizer Investigational Site, Vráble
  - Pfizer Investigational Site, Zvolen

RESULTS

PARTICIPANT FLOW:
Groups:
- Fesoterodine 4 mg or 8 mg: The recommended starting dose was 4 mg once daily. Based upon individual response, the dose was increased to 8 mg once daily.
Period: Overall Study
Arm/Group | Fesoterodine 4 mg or 8 mg
Started | 823
Completed | 816
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1
Not completed — Ongoing at Date of Cut-Off | 4

BASELINE CHARACTERISTICS:
Groups:
- Fesoterodine 4 mg: The recommended starting dose was 4 mg once daily. Based upon individual response, the dose was increased to 8 mg once daily.
Arm/Group | Fesoterodine 4 mg
Number analyzed (Participants) | 823
Age, Customized [Number; unit: participants]
  <18 years | 11
  18-44 years | 102
  44-64 | 497
  >=65 years | 213
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 574
  Male | 249

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Micturition Frequency Per 24 Hours at Each Visit
Description: Micturition frequency: mean number of 'day time' (i.e., the time the participant was awake) micturitions per 24 hours and calculated as the total number of 'day time' urinations, divided by the total diary days collected at that visit.
Time Frame: Baseline, Month 1, Month 2, Month 3 or Early Termination (ET)
Population: The full analysis set (FAS) included all patients who received at least one dose of the study medication and who had at least one post baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Increase of Dose From 4 mg to 8 mg Due to Lack of Efficacy
Number analyzed (Participants) | 754 | 11 | 57
episodes
  Baseline | 11.661 (2.8565) | 10.636 (3.4269) | 12.664 (2.7612)
  Visit 2 (Month 1) | -2.306 (1.5773) | -2.303 (1.2863) | -1.566 (1.4241)
  Visit 3 (Month 2) | -3.482 (1.9022) | -2.848 (1.1772) | -3.160 (1.7571)
  Visit 4 (Month 3 or ET) | -4.180 (2.1018) | -4.000 (1.2293) | -4.031 (1.8995)

2. Secondary Outcome: Change From Baseline in Post Void Residual (PVR) Urine Volume at Visit 2, Visit 3, and Visit 4
Description: The PVR urine volume: measured by an ultrasound scan.
Time Frame: Baseline, Month 1, Month 2, Month 3 or ET
Population: FAS
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Increase of Dose From 4 mg to 8 mg Due to Lack of Efficacy
Number analyzed (Participants) | 754 | 11 | 57
ml
  Baseline | 27.932 (27.6079) | 42.000 (35.6059) | 24.867 (27.7108)
  Visit 2 (Month 1) | -6.650 (16.4784) | -12.800 (13.2313) | -2.364 (11.2500)
  Visit 3 (Month 2) | -9.864 (20.2348) | -18.700 (22.2663) | -5.791 (17.8493)
  Visit 4 (Month 3 or ET) | -12.800 (23.9575) | -21.000 (24.3584) | -7.415 (21.7658)

3. Secondary Outcome: Patient's Global Evaluation of Fesoterodine
Description: The patients global evaluation of study medication was assessed via the question 'how would you rate your overall response to the study medication?' and was assessed on the four point categorical scale, ranging from 'Poor' to 'Excellent'.
Time Frame: Baseline, Month 3 or ET
Population: The safety analysis set (SAS) included all subjects who enrolled in the study, signed informed consent and received at least one dose of study medication.
Measure: Number; unit: participants
Groups:
- All Subjects: Fesoterodine 4 or 8 mg
Arm/Group | All Subjects
Number analyzed (Participants) | 823
participants
  Excellent | 536
  Good | 252
  Fair | 22
  Poor | 10
  Missing | 3

4. Secondary Outcome: Clinical Global Evaluation of Fesoterodine
Description: Clinical global evaluation of study medication was assessed via the question 'how would you rate the study medication the patient received for overactive bladder?,' and was assessed on the four point categorical scale, ranging from 'Poor' to 'Excellent.'
Time Frame: 12 weeks
Population: SAS
Measure: Number; unit: participants
Groups:
- All Subjects: The recommended starting dose was 4 mg once daily. Based upon individual response, the dose was increased to 8 mg once daily.
Arm/Group | All Subjects
Number analyzed (Participants) | 823
participants
  Excellent | 513
  Good | 274
  Fair | 24
  Poor | 9
  Missing | 3

5. Secondary Outcome: Efficacy and Tolerability Compared to Previous Medication (Overall Treatment Effect Scale) at Visit 4
Description: Overall Treatment Effect Scale: 3 questions from which a numeric score was derived. If a subject answered '(2) About the same' to question 1 then a score of 0 was given. If a subject answered '(1) Worse' to question 1, then a score between -7=a very great deal worse to -1=Almost the same, hardly worse at all was given depending on severity of their symptoms (determined from answer to question 2). If a subject answered '(3) Better' to question 1, then a score ranging from 1=Almost the same, hardly better at all to 7=A very great deal better, depending on their answer to question 3, was given.
Time Frame: Month 3 or ET
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Increase of Dose From 4 mg to 8 mg Due to Lack of Efficacy
Number analyzed (Participants) | 754 | 11 | 57
scores on a scale | 5.661 (1.1663) | 5.818 (0.9816) | 4.702 (1.7925)

6. Secondary Outcome: Overactive Bladder Questionnaire (OAB-q): Symptom Severity/Bother Scale
Description: Symptom severity/bother score: sub-section of the OAB-q consists of 8 questions. Each item assessed on ordinal scale (0=Not at all to 5=a very great deal). Score=sum of scores for items 1 to 8 and a further 2 points were added if subject was male. Lowest possible score=0 and highest=42. Data were transformed onto a 0 to 100 scale and analyzed based on the transformed score: Transformed Symptom Bother Score=[(Actual Total Raw Score minus Lowest possible value of raw score) divided by Range] multiplied by 100. Higher scores=greater symptom severity or bother and lower=minimal symptom severity.
Time Frame: Baseline, Month 3 or ET
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Increase of Dose From 4 mg to 8 mg Due to Lack of Efficacy
Number analyzed (Participants) | 754 | 11 | 57
scores on a scale
  Baseline | 59.263 (17.5239) | 70.000 (10.1242) | 64.737 (17.1696)
  Visit 4 (Month 3 or ET) | 25.147 (14.3690) | 35.682 (12.7520) | 32.719 (17.9115)

7. Primary Outcome: Change From Baseline in Nocturnal Micturition Frequency Per 24 Hours at Visit 2, Visit 3, and Visit 4
Description: Nocturnal frequency: mean number of 'night time' (the time the participant was asleep and the urge to urinate woke him/her up) micturitions and calculated as the total number of 'night time' urinations, divided by the total diary days collected at that visit.
Time Frame: Baseline, Month 1, Month 2, Month 3 or ET
Population: FAS
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Increase of Dose From 4 mg to 8 mg Due to Lack of Efficacy
Number analyzed (Participants) | 754 | 11 | 57
episodes
  Baseline | 3.027 (1.2593) | 4.000 (1.4220) | 3.528 (1.3452)
  Visit 2 (Month 1) | -1.104 (0.7960) | -1.212 (0.8065) | -0.915 (0.9115)
  Visit 3 (Month 2) | -1.621 (0.9281) | -1.848 (1.1290) | -1.613 (1.0928)
  Visit 4 (Month 3 or ET) | -1.914 (1.0820) | -2.030 (1.3035) | -2.072 (1.0907)

8. Primary Outcome: Change From Baseline in Urgency Episode Frequency (UEF) Per 24 Hours at Visit 2, Visit 3, and Visit 4
Description: UEF: mean number of micturition related urgency episodes per 24 hours and calculated as the total number of 'urgency' urinations (i.e., sudden urges to urinate and problems to delay micturition) divided by 3 (or if data for 3 days were not available, over the total number of diary days collected at that visit).
Time Frame: Baseline, Month 1, Month 2, Month 3 or ET
Population: FAS
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Increase of Dose From 4 mg to 8 mg Due to Lack of Efficacy
Number analyzed (Participants) | 754 | 11 | 57
episodes
  Baseline | 4.412 (2.4355) | 4.697 (1.9914) | 5.587 (3.7759)
  Visit 2 (Month 1) | -1.890 (1.5967) | -1.697 (0.9827) | -1.650 (1.3065)
  Visit 3 (Month 2) | -2.736 (1.9249) | -2.182 (1.4557) | -2.895 (2.6468)
  Visit 4 (Month 3 or ET) | -3.127 (2.0210) | -2.636 (1.7221) | -3.814 (3.0690)

9. Primary Outcome: Change From Baseline in Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Visit 2, Visit 3, and Visit 4
Description: The mean number of UUI episodes: total number of UUI episodes, divided by the total diary days collected at that visit.
Time Frame: Baseline, Month 1, Month 2, Month 3 or ET
Population: FAS
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Increase of Dose From 4 mg to 8 mg Due to Lack of Efficacy
Number analyzed (Participants) | 754 | 11 | 57
episodes
  Baseline | 2.601 (1.7127) | 2.933 (1.2551) | 3.467 (2.4484)
  Visit 2 (Month 1) | -1.209 (1.0891) | -1.067 (1.1738) | -1.190 (1.2532)
  Visit 3 (Month 2) | -1.806 (1.3107) | -1.583 (1.4974) | -1.781 (1.4729)
  Visit 4 (Month 3 or ET) | -2.065 (1.4582) | -1.733 (1.6836) | -2.362 (1.6477)

10. Secondary Outcome: Change From Baseline in Total Scores of OAB-q at Visit 4
Description: as for outcome 6
Time Frame: Baseline, Month 3 or ET
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Increase of Dose From 4 mg to 8 mg Due to Lack of Efficacy
Number analyzed (Participants) | 754 | 11 | 57
scores on a scale | -34.101 (16.0799) | -34.318 (9.4928) | -32.018 (17.7183)

11. Secondary Outcome: Time To Onset Of Treatment Response
Description: Participant's perception of treatment response assessment since the previous visit was noted at each visit. Time to onset of response was calculated in weeks from start of treatment.
Time Frame: Month 1, Month 2, Month 3 or ET
Population: FAS
Measure: Median (Full Range); unit: weeks
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Increase of Dose From 4 mg to 8 mg Due to Lack of Efficacy
Number analyzed (Participants) | 754 | 11 | 57
weeks | 3.0 (1.27) [0 to 10] | 3.0 (1.10) [1 to 4] | 3.0 (2.72) [1 to 13]

12. Secondary Outcome: Study Doses
Description: Number of subjects that changed doses throughout the study period.
Time Frame: Month 3 or ET
Population: SAS
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 823
participants
  Increased | 57
  Stayed the same | 766
  Decreased | 0
  Fluctuated | 0

13. Secondary Outcome: Reasons for Study Treatment Dose Changes
Description: Possible change in the dose and the reasons for the change were collected and documented.
Time Frame: Month 3 or ET
Population: SAS
Measure: Number; unit: participants
Groups:
- All Subjects: Fesoterodine 4 mg or 8 mg
Arm/Group | All Subjects
Number analyzed (Participants) | 823
participants
  Inefectivity, Not Sufficient Effectivity | 22
  Infectivity | 29
  Insufficient (efficiency) effect | 1
  Insufficient response | 1
  Poor overall response | 1
  Missing | 4

ADVERSE EVENTS:
Groups:
- Fesoterodine 4 mg or 8 mg: All Subjects
Arm/Group | Fesoterodine 4 mg or 8 mg
Serious Adverse Events (participants affected / at risk) | 0/823
Other Adverse Events (participants affected / at risk) | 78/823
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4 mg or 8 mg (N=823)
Constipation (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 66
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Adverse event (General disorders) | 2
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.